#### Statistical Analysis Plan

# Effect of Calcipotriol plus Betamethasone Dipropionate Gel on the HPA Axis and Calcium Metabolism in Adolescent Subjects (Aged 12 to 16 Years, 11 months) with Scalp and Body Psoriasis

A phase 2 trial evaluating the safety and efficacy of once daily use of LEO 80185 gel containing calcipotriol 50 mcg/g plus betamethasone 0.5 mg/g (as dipropionate) in adolescent subjects (aged 12 to 16 years, 11 months) with scalp and body psoriasis

An international, multi-centre, prospective, non-controlled, open, single-group, 8-week trial in adolescent subjects (aged 12 to 16 years, 11 months) with scalp and body psoriasis

| LEO Pharma A/S | Trial ID: | LP0076-1017 |
|----------------|-----------|-------------|
| | Date: | 16-Mar-2018 |
| | Version: | 1.0 |

| Trial ID: <b>LP0076-1017</b> | Date: 16-Mar-2018 | Version: 1.0 |
|------------------------------|-------------------|--------------|

# 1 Statistical Analysis Plan Approval

# 1.1 Approval Statement

QC Statistician, Biostata Aps

On behalf of LEO, the Biostatistics Lead and the Medical Lead, are authorised to approve the Statistical Analysis Plan.

The QC statistician has by approving this document confirmed that the statistical information has been subject to statistical quality control.

The following persons have approved this Statistical Analysis Plan using electronic signatures as presented on the last page of this document.

| PPD | |
|------------------|--------------------------------|
| Biostatistics Le | ad, Global Clinical Operations |
| PPD | |
| Medical Lead, I | Medical Sciences and Safety |
| PPD | |

|------------------------------|-------------------|--------------|

# 2 Statistical Analysis Plan Statements

# 2.1 Compliance with Good Clinical Practice

This Statistical Analysis Plan is designed to comply with the standards issued by the International Conference on Harmonisation (ICH) (E3: Structure and Content of Clinical Study Reports, E6: Good Clinical Practice, and E9: Statistical Principles for Clinical Trials).

|------------------------------|-------------------|--------------|

# **Table of Contents**

| 1 Statistical Analysis Plan Approval | 2 |
|------------------------------------------------|----|
| 1.1 Approval Statement | 2 |
| 2 Statistical Analysis Plan Statements | 3 |
| 2.1 Compliance with Good Clinical Practice | 3 |
| Table of Contents | 4 |
| 3 List of Abbreviations | 5 |
| 3.1 List of Abbreviations | 5 |
| 4 Statistical Analysis Plan Authors | 5 |
| 5 Introduction | 5 |
| 6 Statistical Analysis | 7 |
| 6.1 Baseline Considerations | 7 |
| 6.1.1 Compliance | 8 |
| 6.2 Analysis of Efficacy | 9 |
| 6.3 Analysis of Safety | 9 |
| 6.4 ACTH-Challenge | 9 |
| 6.4.1 Exposure | 10 |
| 6.4.2 Drug Accountability | 10 |
| 6.4.3 Adverse Events | 11 |
| 6.4.4 Laboratory Data | 12 |
| 6.4.5 Other observations | 12 |
| 6.5 General Principles | 13 |
| 6.5.1 Pooling of Trial Sites | 13 |
| 6.5.2 Handling of Drop-outs and Missing Values | 13 |
| 6.5.4 Treatment Labels | 15 |
| Annendix I | 16 |

|------------------------------|-------------------|--------------|

#### 3 List of Abbreviations

#### 3.1 List of Abbreviations

ACTH Adrenocorticotropic hormone

AE Adverse Event
CRF Case Report Form
CTR Clinical Trial Report

ICH International Conference on Harmonisation

IGA Investigator's global assessment
LOCF Last Observation Carried Forward
LLOQ Lower Limit of Quantification
IMP Investigational Medicinal Product

MedDRA Medical Dictionary for Regulatory Activities

PASI Psoriasis Area and Severity Index

PK Pharmacokinetics

SAP Statistical Analysis Plan

#### 4 Statistical Analysis Plan Authors

PPD , MSc, Senior Statistician, Biostatistics, LEO Pharma A/S, DK-2750, Ballerup, Denmark, tel: +45 PPD , e-mail: PPD @leo-pharma.com

PPD , MSc, Senior Statistician, Biostatistics, LEO Pharma A/S, DK-2750, Ballerup, Denmark, tel: +45 PPD @leo-pharma.com

PPD , PhD, Clincal Project Manager, Trial Management, LEO Pharma A/S, DK-2750, Ballerup, Denmark, tel: +45 PPD , e-mail: PPD @leo-pharma.com

PPD , MSc, Principal Medical Writer, Medical Communication, LEO Pharma A/S, DK-2750, Ballerup, Denmark, tel: +45 PPD , e-mail: PPD @leo-pharma.com

PPD , MD PhD, Principal Medical Expert, Medical Department, LEO Pharma A/S, DK-2750, Ballerup, Denmark, tel: +45 PPD , e-mail: PPD @leo-pharma.com

#### 5 Introduction

The statistical analysis will be performed as outlined in the Consolidated Clinical Study Protocol. This Statistical Analysis Plan, prepared after review of the data, contains a more technical and detailed elaboration of some points in the statistical analysis described in the

|------------------------------|-------------------|--------------|

protocol. Minor deviations from the planned data presentation and analysis are accounted for. The analysis sets which are to be used for the statistical analysis are presented in Analysis Set Definition Document.

Table 1 includes protocol amendments that are relevant to the statistical reporting. The inclusion criteria for subjects *not* performed HPA and PK assessments has been updated in Consolidated Clinical Study Protocol, version 4.0, dated 16-Feb-2015. The extent of psoriasis required on the body and the severity of psoriasis required on the body and the scalp has been revised to better reflect psoriasis commonly seen in the adolescent population. The definition of 'controlled disease' under the secondary response criteria was updated accordingly. More details can be found in LP0076-1017 Summary of Amendment(s) to a Clinical Trial Authorisation, 02-Mar-2015 (v1.0).

Table 1: Protocol amendments that are relevant to the statistical reporting.

| Section no in Consolidated | То | From: |
|---|---|---|
| Clinical Study Protocol | | |
| version 4.0 and 6.0 | | |
| 10.4.1.3 (a and b, BODY) | At SV2 and Visit 1, a clinical | At SV2 and Visit 1, a clinical |
| | diagnosis of body (trunk and/or | diagnosis of scalp and body (trunk |
| The inclusion criteria for subjects | limbs) psoriasis which is: | and/or limbs) psoriasis which is: |
| not performing HPA and PK assessments was updated. | a. more than or equal to 3% of the | a. of an extent of 10 to 35% of the |
| assessments was updated. | body surface area (excluding | body surface area (excluding |
| | psoriatic lesions of the face and | psoriatic lesions of the face and |
| | sensitive areas), and | sensitive areas. Sensitive areas |
| | b. of at least <i>mild</i> severity | include armpits, groin, under the |
| | according to the investigator's | breasts and in other skin folds |
| | global assessment of disease | around the genitals and buttocks), |
| | severity on the body. | and |
| | At SV2 and Visit 1, a clinical | b. of at least <i>moderate</i> severity |
| | diagnosis of scalp psoriasis which | according to the investigator's |
| | is: | global assessment of disease |
| | a. more than or equal to 10% of the | severity on the body. |
| | scalp area, and | |
| | - | |
| | b. of at least mild severity | |
| | according to the investigator's | |
| | global assessment of disease | |
| | severity on the scalp | |

|------------------------------|-------------------|--------------|

| 10.4.1.3 (a and b, SCALP) | At SV2 and Visit 1, a clinical | At SV2 and Visit 1, a clinical |
|---|---|---|
| | diagnosis of scalp psoriasis which | diagnosis of scalp psoriasis which |
| The inclusion criteria for subjects | is: | is: |
| not performing HPA and PK assessments was updated. | a. more than or equal to 10% of the scalp area, and | a. more than or equal to 10% of the scalp area, and |
| | b. of at <b>least mild</b> severity | b. of at least <i>moderate</i> severity |
| | according to the investigator's | according to the investigator's |
| | global assessment of disease | global assessment of disease |
| | severity on the scalp | severity on the scalp. |
| | , . | _ |
| 10.10.1 | Subjects with "Controlled disease" | Subjects with "Controlled disease" |
| | (i.e., "Clear" or "Almost clear" for | (i.e., "Clear" or "Almost clear") |
| Revised secondary response | subjects with at | according to the investigator's |
| criteria. | least "Moderate" disease at | global assessment of disease |
| | baseline, "Clear" for subjects with | severity on the body at end of |
| | "Mild" disease at baseline) | treatment. |
| | according to the investigator's | |
| | global assessment of disease | |
| | severity on the body at | |
| | end of treatment. | |

# 6 Statistical Analysis

The statistical analysis will be carried out as described in the Consolidated Clinical Study Protocol with a few exceptions as described below.

Lists of planned tables, figures and individual subject data listings for the Clinical Trial Report are provided in Appendix 1.

#### **6.1 Baseline Considerations**

According to the protocol descriptive statistics of demographics and other baseline characteristics will be presented for all subjects in the safety analysis set and per protocol analysis set as these are the datasets used for primary response criteria.

Age and sex will be presented by country and not by centre as described in the protocol, due to too few number of subjects at most centres.

The age will be presented in three categories:

|------------------------------|-------------------|--------------|

- Overall
- 12 to 14 years
- 15 to <17 years.

A table of serum cortisol concentrations at time 0, and at 30 and 60 min after ACTH challenge at baseline, although not planned in the protocol, will be produced for the per protocol analysis set.

Any abnormalities recorded during physical examination will be included in concurrent diagnoses table.

The baseline is defined as last assessment performed prior the first application of IMP.

#### 6.1.1 Compliance

As described in the protocol, compliance with treatment instructions will be tabulated for all subjects who applied any IMP. Compliance with treatment instructions will be presented for all subjects in the safety analysis set and per protocol analysis set. Compliance is defined by number of missed days due to other reasons than cleared psoriasis in relation to treatment period. Treatment period is defined as the number of days from the treatment assignment at Visit 1 to either trial completion or early withdrawal.

The number and percentage of subjects who either did or did not comply with the trial treatment regimen will be summarized. The extent of non-compliance as categories of the percentage of applications missed will also be presented:

- No
- Yes: <=10% applications missed
- Yes: >10% to <=20% applications missed
- Yes: >20% to <=30% applications missed
- Yes: >30% to <=40% applications missed
- Yes: >40% to <=50% applications missed
- Yes: >50% applications missed
- Total

|------------------------------|-------------------|--------------|

#### **6.2** Analysis of Efficacy

The statistical analysis of efficacy will be based on the full analysis set according to the defined response criteria in the protocol.

'Controlled disease' will be presented in a table by age group, the categories to be used are the same as defined in section 6.1.

Additional tables, not planned in the protocol, will be produced:

- Controlled disease (IGA on the body) at end of treatment by race
- Controlled disease (IGA on the body) at end of treatment by baseline total extent of psoriasis

Baseline for the efficacy is defined as last observation collected prior the first application of IMP, and is defined as Visit 1 for all assessments.

#### 6.3 Analysis of Safety

The analysis of safety will be based on the safety analysis set according to the defined response criteria in the protocol, with the exception of the ACTH-challenge test which will be based on the per protocol analysis set.

Baseline for the safety analysis is defined as last observation collected prior the first application of IMP, which is Screening Visit 2.

# 6.4 ACTH-Challenge

The results from the ACTH-challenge will be presented as described in the protocol for the per protocol analysis set.

According to the ACTH-challenge procedure described in the protocol, samples of venous blood were to drawn exactly 30 min and 60 min after the CORTROSYN®/SYNACTHIEN® injection, however a time deviation of +/- 10 minutes is considered acceptable as the overall value of the test is to observe substantial increases in cortisol levels and identify adrenal insufficiency up to 1 hour after the initial injection, therefore the exact timing of the incremental time points (30 and 60 minutes) is of less importance. Samples outside the acceptable deviation will not be included in the analysis. No measurements outside the acceptable deviation were observed.

|------------------------------|-------------------|---------------|

#### 6.4.1 Exposure

As described in the protocol, the duration of exposure (weeks) and extent of exposure (subject-treatment-weeks) to LEO 80185 will be summarized for the safety analysis set.

#### 6.4.2 Drug Accountability

The amount of IMP used in grams and the average weekly amount used in grams will be tabulated for the safety analysis set, and separately for three different treatment periods (first four weeks, second four weeks, and the total treatment period).

The average weekly amount of IMP used, during the total treatment period, in defined usage categories, will be tabulated; this table was not planned in the protocol:

- <20 g/week
- 20 to <40 g/week
- >=60 g/week
- Total

The mean weight of full bottles, including label of IMP, is presented in Table 1 for each batch and kit number. Also the label type is given.

Table 2: Mean weight of full bottles of IMP by batch number and kit number

| Batch number | Kit number | Weight of a full bottle + label (g) | Label Type |
|---|---|---|---|
| 131537101 | 0001 - 3200 | 86.8 g | Booklet |
| P14090 | 3201 - 4757 | 86.9 g | Booklet |
| P14090 | 4758 - 5600 | 86.6 g | Single panel |
| P14090 | 5797-5955 | 87.0 g | Single panel |

For each treatment period the following rules for calculating amount of IMP used will apply.

For each subject the weight of IMP used for a particular treatment period will be determined by calculating the difference between the weight of a set of full bottles dispensed and the weight of the returned bottles.

If any subjects received bottles for a particular treatment period but did not return them all, then the amount of IMP used for that treatment period will not be calculated. If any bottles are

|------------------------------|-------------------|---------------|

not dispensed, they will not contribute to the weight of IMP used for that treatment period. If any bottles are returned with their seal unbroken, the weight of IMP used from that bottle will be assigned a value of zero. If a returned bottle weighs more than the estimated mean weight of a full bottle, it will be assumed that zero grams were used.

The average weekly amount of IMP used will be calculated for each subject as the amount of IMP used for a particular treatment period, divided by the duration (days) of the treatment period and then multiplied by 7.

#### **6.4.3** Adverse Events

The AEs will be presented for the safety analysis set as described in the protocol.

The AEs are coded in accordance with the MedDRA dictionary version 15.1.

The number of events will be presented in all adverse events tables where number of subjects is presented.

One subject had a serious adverse event and one subject was withdrawn early from the trial due to an adverse event, therefore serious adverse events and adverse events leading to withdrawal will not be tabulated, but will be evaluated separately in the report.

Additional tables, not planned in the protocol will be produced:

- Adverse events by age group, MedDRA, primary system organ class and preferred term
- Adverse events by sex, MedDRA primary system organ class and preferred term
- Adverse events by race, MedDRA primary system organ class and preferred term
- Adverse events by baseline IGA on the body, MedDRA primary system organ class and preferred term
- Adverse events by baseline total extent of psoriasis, MedDRA primary system organ class and preferred term
- Adverse events by IMP usage (<40 g/week, ≥40 g/week), MedDRA primary system organ class and preferred term.

Adverse events will be presented separately for subjects using at least 40 g per week of IMP during the total treatment period and for those using less than 40 g per week of IMP during the total treatment period.

|------------------------------|-------------------|---------------|

## 6.4.4 Laboratory Data

The laboratory data will be presented for the safety analysis set as described in the protocol.

However, 25-hydroxy vitamin D baseline values will not be summarized since no abnormal values have been observed.

The following approach will be used in case of repeated or missed laboratory measurements:

- if an initial measurement was normal but the measurement was still repeated then the initial measurement will be presented in the tables and both measurements will be included in the listing.
- if an initial measurement was repeated by mistake then the initial measurement will be presented in the tables and both measurements will be included in the listing.
- if an initial measurement was abnormal and the measurement was repeated due to a technical problem then the repeated measurement will be presented in the tables and both measurements will be included in the listing.
- if an initial measurement was missing but a measurement from an unscheduled visit is available and the unscheduled visit was performed within 5 days after the actual visit then the measurement from the unscheduled visit will be used, for example one measurement from an unscheduled visit after Visit 3 will be included in the analysis of albumin corrected serum calcium (gives a total of 100 measurements).

The number of measurements outside the reference range will be presented in relevant laboratory tables. The number of measurements for other than primary and secondary endpoints that fall outside the limit for quantification will be presented in relevant laboratory tables.

#### 6.4.5 Other observations

#### PK evaluation

As most plasma concentrations were below LLOQ the PK parameters will not be calculated at Week 4 for each assayed compound.

Plasma concentrations will be presented in the listing.

#### Vital signs

|------------------------------|-------------------|---------------|

For systolic and diastolic blood pressure and heart rate, the absolute value by visit and change from baseline (SV2) to Week 4 (Visit 3) and Week 8 (Visit 5) will be summarized

Clinically significant abnormalities in the vital signs at baseline (SV2), Week 4 and/or Week 8 will not be presented since no clinically significant abnormalities were observed. Any abnormalities at Week 4 and/or Week 8 that were not present at baseline will be presented in the listing.

The following approach will be used in case of repeated vital signs measurements:

- if an initial measurement was normal but the measurement was still repeated then the initial measurement will be presented in the tables
- if an initial measurement was abnormal and the measurement was repeated then the average of both measurements will be presented in the tables.

All measurements will be included in the listings (initial measurement and repeated measurements).

#### 6.5 General Principles

## 6.5.1 Pooling of Trial Sites

There will be no pooling of centres.

# 6.5.2 Handling of Drop-outs and Missing Values

The efficacy and laboratory data will be tabulated by visit using an observed cases approach except for the tabulation of end of treatment values for which the LOCF approach will be used.

The extent of missing values are described in

|------------------------------|-------------------|---------------|

Table 3 for the primary endpoints and secondary endpoints involving laboratory measurements:

|------------------------------|-------------------|---------------|

Table 3: Number of missing values and number of observations/Total.<sup>1</sup>

| | Number of Missing Values | | | |
|---|---|---|---|---|
| | (Number of observations/Total) | | | otal) |
| Endpoint | Test | Screening Visit 2 | Week 4 | Week 8 |
| Primary | Albumin corrected | 0 | 5 | 3 |
| Filliary | serum calcium | (107/107) | (99/104) | (87/90) |
| Duino aut | 24-hours urinary | 9 | 12 | 11 |
| Primary | calcium excretion | (98/107) | (92/104) | (79/90) |
| Duino aut | Serum Cortisol at | 0 | 1 | 1 |
| Primary | time 0 | (33/33) | (31/32) | (29/30) |
| Deimory | Serum Cortisol at | 0 | 1 | 1 |
| Primary | time 30 min <sup>2</sup> | (33/33) | (31/32) | (29/30) |
| Duine | Serum Cortisol at | 0 | 1 | 1 |
| Primary | time 60 min <sup>2</sup> | (33/33) | (31/32) | (29/30) |
| | Urinary | 9 | 12 | 11 |
| Secondary | calcium:creatinine | - | | |
| | ratio | (98/107) | (92/104) | (79/90) |
| Caran James | Serum alkaline | 0 | 5 | 3 |
| Secondary | phosphatase | (107/107) | (99/104) | (87/90) |

<sup>1:</sup> Duplicates by subject, visit and numerical results are excluded. The table includes only subjects assigned to treatment

<sup>2:</sup> Serum Cortiosol 30 min and 60 min after ACTH challenge

|------------------------------|-------------------|---------------|

# **6.5.4** Treatment Labels

The treatment label to be used in text and tables in the CTR and in the individual subject data listings is 'LEO 80185'.

|------------------------------|-------------------|---------------|

# Appendix I

Tables, Figures and Listings

|------------------------------|-------------------|---------------|

# **Tables and Figures, Baseline Characteristics and Investigational Product Data (Module 2)**

#### **Tables**

- Table 1-1 Subject enrolment and treatment assignment by country and by centre: enrolled subjects and subjects assigned treatment
- Table 1-2 Reasons for withdrawal during the screening phase: enrolled subjects.
- Table 1-3 Reasons for withdrawal during the treatment phase: safety analysis set and per protocol analysis set
- Table 1-4 Sex, ethnicity, race and skin type: safety analysis set and per protocol analysis set
- Table 1-5 Age, BMI, height, weight and duration of psoriasis: safety analysis set and per protocol analysis set
- Table 1-6 Investigator's global assessment of disease severity on the body at baseline: safety analysis set and per protocol analysis set
- Table 1-7 Patient's global assessment of disease severity on the body at baseline: safety analysis set and per protocol analysis set
- Table 1-8 Investigator's assessment of extent of psoriasis at baseline: safety analysis set and per protocol analysis set
- Table 1-9 PASI at baseline: safety analysis set and per protocol analysis set
- Table 1-10 Concomitant medication at baseline: safety analysis set and per protocol analysis set
- Table 1-11 Concurrent diagnoses at baseline: safety analysis set and per protocol analysis set
- Table 1-12 Age by country: safety analysis set and per protocol analysis set
- Table 1-13 Sex by country: safety analysis set and per protocol analysis set
- Table 1-14 Serum cortisol concentration at time 0, and at 30 and 60 min after ACTH challenge at baseline: per protocol analysis set

|------------------------------|-------------------|---------------|

Table 1-15 Compliance with treatment instructions: safety analysis set and per protocol analysis set

#### **Figures**

Figure 1-1 Visit attendance: enrolled subjects Figure 1-2 Trial analysis sets: enrolled subjects

#### Tables and Figures, Efficacy Data (Module 3)

#### **Tables**

Table 2-1 Investigator's global assessment of disease severity on the body by visit and at end of treatment: full analysis set

Table 2-2 Controlled disease (IGA on the body) by visit and at end of treatment: full analysis set

Table 2-3 Controlled disease (IGA on the body) at end of treatment by age group: full analysis set

Table 2-4 Controlled disease (IGA on the body) at end of treatment by sex: full analysis set

Table2-5 Controlled disease (IGA on the body) at end of treatment by race: full analysis set

Table 2-6 Controlled disease (IGA on the body) at end of treatment by baseline IGA on the body: full analysis set

Table 2-7 Controlled disease (IGA on the body) at end of treatment by baseline total extent of psoriasis: full analysis set

Table 2-8 Controlled disease (IGA on the body) at end of treatment by country: full analysis set

Table 2-9 PASI by visit and at end of treatment: full analysis set

Table 2-10 Percentage change in PASI from baseline to each visit and end of treatment: full analysis set

|------------------------------|-------------------|---------------|

- Table 2-11 Investigator's global assessment of disease severity on the scalp by visit and at end of treatment: full analysis set
- Table 2-12 Controlled disease (IGA on the scalp) by visit and at end of treatment: full analysis set
- Table 2-13 Investigator's assessment of extent of psoriasis (total involvement as % of BSA) at baseline, Week 4 and Week 8: full analysis set and per protocol analysis set
- Table 2-14 Investigator's assessment of extent of psoriasis (on body as % of BSA) at baseline, Week 4 and Week 8: full analysis set and per protocol analysis set
- Table 2-15 Investigator's assessment of extent of psoriasis (on scalp as % of scalp area) at baseline, Week 4 and Week 8: full analysis set and per protocol analysis set
- Table 2-16 Patient's global assessment of disease severity on the body by visit and at end of treatment: full analysis set
- Table 2-17 Controlled disease (patient's global assessment on the body) by visit and at end of treatment: full analysis set
- Table 2-18 Patient's global assessment of disease severity on the scalp by visit and at end of treatment: full analysis set
- Table 2-19 Controlled disease (patient's global assessment on the scalp) by visit and at end of treatment: full analysis set
- Table 2-20 Patient's assessment of itching on the body by visit and at end of treatment: full analysis set
- Table 2-21 Change in itching on the body from baseline to each visit and at end of treatment: full analysis set
- Table 2-22 Patient's assessment of itching on the scalp by visit and at end of treatment: full analysis set
- Table 2-23 Change in itching on the scalp from baseline to each visit and at end of treatment: full analysis set
- Table 2-24 Patient's assessment of sleep loss by visit and at end of treatment: full analysis set

|------------------------------|-------------------|---------------|

Table 2-25 Change in sleep loss from baseline to each visit and end of treatment: full analysis set

#### **Tables and Figures, Safety Data (Module 4)**

#### **Tables**

Table 3-1 Subjects with serum cortisol concentration <=18 mcg/dL at 30 minutes after ACTH challenge at Week 4 and Week 8: per protocol analysis set

Table 3-2 Subjects with serum cortisol concentration <=18 mcg/dL at both 30 and 60 minutes after ACTH challenge at Week 4 and Week 8: per protocol analysis set

Table 3-3 Serum cortisol concentration at time 0 and at 30 and 60 minutes after ACTH challenge at baseline, Week 4 and Week 8: per protocol analysis set

Table 3-4 Individual data for subjects with serum cortisol concentration <=18 mcg/dL at either 30 minutes or 60 minutes after ACTH challenge: per protocol analysis set

Table 3-5 Change in albumin-corrected serum calcium from baseline to Week 4, Week 8 and end of treatment: safety analysis set

Table 3-6 Albumin-corrected serum calcium at baseline, Week 4, Week 8 and end of treatment: safety analysis set

Table 3-7 Albumin-corrected serum calcium categorised as low, normal or high at Week 4, Week 8 and end of treatment shown against baseline category: safety analysis set

Table 3-8 Change in 24-hour urinary calcium excretion from baseline to Week 4, Week 8 and end of treatment: safety analysis set

Table 3-9 24-hour urinary calcium excretion at baseline, Week 4, Week 8 and end of treatment: safety analysis set

Table 3-10 24-hour urinary calcium excretion categorised as low, normal or high at Week 4, Week 8 and end of treatment shown against baseline category: safety analysis set

Table 3-11 Change in 24-hour urinary calcium excretion from baseline to Week 4, Week 8 and end of treatment in subjects with complete urinary collection: safety analysis set

|------------------------------|-------------------|---------------|

- Table 3-12 24-hour urinary calcium excretion at baseline, Week 4, Week 8 and end of treatment in subjects with complete urinary collection: safety analysis set
- Table 3-13 24-hour urinary calcium excretion categorised as low, normal or high at Week 4, Week 8 and end of treatment shown against baseline category in subjects with complete urinary collection: safety analysis set
- Table 3-14 Change in urinary calcium:creatinine ratio from baseline to Week 4 and Week 8: safety analysis set
- Table 3-15 Urinary calcium:creatinine ratio categorised as low, normal or high at Week 4 and Week 8 shown against baseline category: safety analysis set
- Table 3-16 Change in serum alkaline phosphatase from baseline to Week 4 and Week 8: safety analysis set
- Table 3-17 Serum alkaline phosphatase categorised as low, normal or high at Week 4 and Week 8 shown against baseline category: safety analysis set
- Table 3-18 Change in haematology parameters from baseline to Week 4 and Week 8: safety analysis set
- Table 3-19 Change in other biochemistry parameters from baseline to Week 4 and Week 8: safety analysis set
- Table 3-20 Change in other urinalysis parameters from baseline to Week 4 and Week 8: safety analysis set
- Table 3-21 Haematology parameters at baseline, Week 4 and Week 8: safety analysis set
- Table 3-22 Haematology parameters categorised as low, normal or high at Week 4 and Week 8 shown against baseline category: safety analysis set
- Table 3-23 Biochemistry parameters at baseline, Week 4 and Week 8: safety analysis set
- Table 3-24 Other biochemistry parameters categorised as low, normal or high at Week 4 and Week 8 shown against baseline category: safety analysis set
- Table 3-25 Urinalysis parameters at baseline, Week 4 and Week 8: safety analysis set

|------------------------------|-------------------|---------------|

Table 3-26 Other urinalysis parameters categorised as low, normal or high at Week 4 and Week 8 shown against baseline category: safety analysis set

Table 3-27 Presence of urinary glucose and ketones at Week 4 and Week 8 against presence at baseline: safety analysis set

Table 3-28 Duration and extent of exposure to treatment: safety analysis set

Table 3-29 Amount of IMP used: safety analysis set

Table 3-30 Average weekly amount of IMP used: safety analysis set

Table 3-31 Average weekly amount of IMP used in defined usage categories: safety analysis set

Table 3-32 Overall summary of adverse events: safety analysis set

Table 3-33 Adverse events by MedDRA primary system organ class: safety analysis set

Table 3-34 Adverse events by MedDRA primary system organ class and preferred term: safety analysis set

Table 3-35 Intensity of adverse events by MedDRA primary system organ class and preferred term: safety analysis set

Table 3-36 Causal relationship of adverse events to IMP by MedDRA primary system organ class and preferred term: safety analysis set

Table 3-37 Adverse drug reactions by MedDRA primary system organ class and preferred term: safety analysis set

Table 3-38 Intensity of adverse drug reactions by MedDRA primary system organ class and preferred term: safety analysis set

Table 3-39 Lesional/perilesional adverse events by MedDRA primary system organ class and preferred term: safety analysis set

Table 3-40 Lesional/perilesional adverse events on the body by MedDRA primary system organ class and preferred term: safety analysis set

|------------------------------|-------------------|---------------|

Table 3-41 Lesional/perilesional adverse events on the scalp by MedDRA primary system organ class and preferred term: safety analysis set

Table 3-42 Adverse events by age group, MedDRA primary system organ class and preferred term: safety analysis set

Table 3-43 Adverse events by sex, MedDRA primary system organ class and preferred term: safety analysis set

Table 3-44 Adverse events by race, MedDRA primary system organ class and preferred term: safety analysis set

Table 3-45 Adverse events by baseline IGA on the body, MedDRA primary system organ class and preferred term: safety analysis set

Table 3-46 Adverse events by baseline total extent of psoriasis, MedDRA primary system organ class and preferred term: safety analysis set

Table 3-47 Adverse events by IMP usage (<40 g/week, ≥40 g/week), MedDRA primary system organ class and preferred term: safety analysis set

Table 3-48 Systolic blood pressure by visit: safety analysis set

Table 3-49 Change in systolic blood pressure from baseline to Week 4 and Week 8: safety analysis set

Table 3-50 Diastolic blood pressure by visit: safety analysis set

Table 3-51 Change in diastolic blood pressure from baseline to Week 4 and Week 8: safety analysis set

Table 3-52 Heart rate by visit: safety analysis set

Table 3-53 Change in heart rate from baseline to Week 4 and Week 8: safety analysis set

|------------------------------|-------------------|---------------|

#### **Patient Data Listings (Appendix 1)**

1-7 Subjects Receiving Investigational Product from Specific Batches

### **Patient Data Listings (Appendix 2)**

Appendix 2.1: Discontinued Subjects

Listing 1-1 Screening Failures

Listing 1-2 Reason(s) for Withdrawal from Trial

Appendix 2.2: Protocol Deviations

Listing 2-1 Protocol Deviations

Listing 2-2 Comments from CRF

Appendix 2.3: Trial Analysis Sets

Listing 3-1 Trial Analysis Set

Listing 3-2 Reasons for Exclusion from Analysis Set

Appendix 2.4: Demographic Data

Listing 4-1 Demographics

Listing 4-2 Duration of Psoriasis Vulgaris.

Listing 4-3 Actual Trial Period

Listing 4-4 Medical History

|------------------------------|-------------------|---------------|

Listing 4-5 Concomitant Diagnoses at Baseline

Listing 4-6 Concomitant Medication

Appendix 2.5: Compliance and/or Investigational Product Concentration Data

Listing 5-1 Compliance

Listing 5-2 Drug Accountability

Listing 5-3 Exposure Dates

Appendix 2.6: Efficacy Data

Listing 6-1: Investigator's Global Assessment of Disease Severity

Listing 6-2: Investigator's Assessment of Extent of Psoriasis

Listing 6-3: Investigator's Assessment of Extent and Severity of Clinical Signs and PASI Score

Listing 6-4: Patient's Global Assessment of Disease Severity

Listing 6-5: Patient's Assessment of Itch and Sleep Loss

Appendix 2.7: Safety Data

Listing 7-1 Deaths

Listing 7-2 Serious Adverse Events

Listing 7-3 Subjects withdrawn due to AE

Listing 7-4 Severe Adverse Events

Listing 7-5 Adverse Events

|------------------------------|-------------------|---------------|

Listing 7-6 Dietary Calcium Intake

Appendix 2.8: Listing of Laboratory Values by Subject

Listing 8-1 Physical Examination, Abnormal Findings

Listing 8-2 Laboratory Measurements

Listing 8-3 Abnormal Laboratory Measurements

Listing 8-4 Vital Signs

Listing 8-5 ACTH Challenge Test

Listing 8-6 Plasma Concentrations.

#### Additional Tables for Results Reporting in Clinical Trial Data Registries

Table 4-1 Age group: subjects assigned to treatment

Table 4-2 Non-serious AEs occurring in ≥[X]% subjects by MedDRA primary SOC and

preferred term: safety analysis set

[Note: X% is 5% or smaller percentage]

# Signature Page for TMF-000048500 v1.0

| Reason for signing: Approved | Approver Verdict(s) Name: PPD Capacity: Biostatistics Date of signature: 16-Mar-2018 10:08:46 GMT+0000 |
|---|---|
| Reason for signing: Approved | Management / Lead Approver Verdict(s) Name: PPD Capacity: Biostatistics Date of signature: 16-Mar-2018 10:56:20 GMT+0000 |
| Reason for signing: Approved | Management / Lead Approver Verdict(s) Name: PPD Capacity: Medical Date of signature: 16-Mar-2018 15:23:52 GMT+0000 |

Signature Page for TMF-000048500 v1.0